CLINICAL TRIAL: NCT05951049
Title: A Phase 2, Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of AT-02
Brief Title: A Study of AT-02 in Subjects With Systemic Amyloidosis.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Attralus, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT02-003
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Amyloidosis; Systemic
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- A (AT-02) (Experimental): Subjects will receive AT-02 via intravenous infusion once every two or 4 weeks for 104 weeks (52 total AT-02 administrations).
  Interventions: Drug: AT02

INTERVENTIONS:
Drug: AT02 — Dosage Form: Solution for injection/infusion Dosage level: Different dose levels of AT02 Route of Administration: Intravenous use

SUMMARY:
This is a Phase 2 open-label extension study to evaluate the long-term safety, tolerability, and clinical activity of AT-02.

AT-02 is an investigational medicinal product being developed to treat systemic amyloidosis.

DETAILED DESCRIPTION:
The study will enroll subjects with systemic amyloidosis who have participated in AT02-001 study and will also directly enroll AL participants with renal disease who did not participate in study AT02-001.

The study includes screening period (56 days), treatment period (week 104), follow up (week 112).

The total duration of participant in study is up to 120 weeks.

A Safety Review Committee (SRC) will periodically convene and review all available clinical and laboratory data during the study. A single SRC will monitor safety across all AT-02 studies to ensure that safety signals are assessed in aggregate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands the study procedures and can give signed informed consent.
2. Subject is willing and able to comply with this protocol and will be available for the entire duration of the study.
3. Has a confirmed diagnosis of AL amyloidosis and meets the criteria below:

   1. Histologic confirmation with a biopsy containing deposits of apple-green birefringent, Congophilic material or other amyloid staining (i.e., thioflavin T or sulfated alcian blue) with confirmatory immunohistochemistry or mass spectrometry, AND
   2. May be receiving maintenance daratumumab and must have achieved and maintained a hematologic very good partial response (VGPR) or complete response (CR), have completed chemotherapy therapy (ie, melphalan, bortezomib, thalidomide, lenalidomide, or cyclophosphamide) and be at least 6 months from first hematologic response (CR or VGPR), AND
   3. Either

   <!-- -->

   1. Screening eGFR ≥20 and ≤75 mL/min/1.73m2 based on CKD-EPI equation, OR
   2. Proteinuria that is not improving (e.g., <25% reduction in urine protein creatinine ratio (UPCR) in the last 12 months or since hematologic response, whichever is shorter) with screening urine albumin creatinine ratio (UACR) >700 mg/g based on central lab assessment of first morning void urine collected at screening and confirmed by a separate Screening 24-hr urine protein >1.0gm/day; 24-hr urine protein may be repeated once during Screening.

   Note: Participants may meet both eGFR and proteinuria criteria
4. Women of childbearing potential (WOCBP):

   1. WOCBP must have a negative serum or urine pregnancy test within 24 hours prior to the start of study treatment.
   2. Must not be breastfeeding, lactating, or planning a pregnancy during the study period.
   3. WOCBP who are not exclusively in same-sex relationships must agree to remain abstinent (complete avoidance of heterosexual intercourse) or use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, during the treatment period and for at least 105 days after the last dose of study intervention.
5. Women of non-childbearing potential (WONCBP), and female participants with vasectomized male partners:

   1. WONCBP must agree to remain abstinent (complete avoidance of intercourse) or the male partners of WONCBP participants must wear a condom to protect against the transfer of study intervention through bodily fluids during the treatment period and for at least 105 days after the last dose of study intervention.
   2. Postmenopausal females must have a documented serum FSH level >40 mIU/mL at Screening to confirm menopause.
6. Male participants:

   1. Male participants must inform their female sexual partners who are WOCBP of the contraceptive requirements of the protocol and are expected to adhere to using contraception with their partner.
   2. Male participants with female sexual partners who are WOCBP must agree to remain abstinent (complete avoidance of heterosexual intercourse) or use adequate contraceptive methods, defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner, during the treatment period and for at least 165 days after the last dose of study intervention.
   3. Male participants must not donate sperm for at least 165 days after the last dose of study intervention.
   4. Male participants in same-sex relationships or in relationships with WONCBP, must agree to remain abstinent (complete avoidance of intercourse) or use a condom to prevent exposure of the partner to study intervention through ejaculate/seminal fluid during the treatment period and for at least 165 days after the last dose of study intervention.

Exclusion Criteria:

1. Receiving hemodialysis or peritoneal dialysis.
2. Myocardial infarction within 3 months of Screening.
3. New York Heart Association Class IV heart failure.
4. Kidney disease not caused by AL amyloidosis.
5. Respiratory insufficiency requiring oxygen therapy.
6. Currently receiving: melphalan, bortezomib, thalidomide, lenalidomide, or cyclophosphamide.
7. Currently receiving unfractionated heparin or heparin analogs (e.g., enoxaparin, dalteparin).
8. Active malignancy with exception of basal cell carcinoma of the skin, curatively resected squamous cell carcinoma of the skin, curatively treated in situ cervical cancer, non-metastatic prostate adenocarcinoma stably managed on hormonal therapy by medical oncologist or for which appropriate management is observation alone.
9. Uncontrolled or active infection.
10. Autoimmune disease requiring treatment with immunosuppressive/modulating treatment in the last year.
11. History of solid organ transplantation.
12. Suspected or known substance abuse disorder(s), serious psychiatric or any other medical condition, which, in the opinion of the Investigator, makes the participant unsuitable.
13. Has any concurrent illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the participant.
14. Screening alanine transaminase (ALT) or aspartate transaminase (AST) is >2.5x upper limit of normal (ULN).
15. Screening estimated creatinine clearance/eGFR using the CKD-EPI equation is <20 mL/min/1.73 m2.
16. Currently participating in an interventional clinical study or has participated in another interventional clinical study within the last four (4) weeks or within five (5) half-lives of the prior study treatment, whichever is longer. This exclusion does not apply to clinical studies in which the only investigational product is a diagnostic agent.
17. Any contraindication to MRI.
18. Hypersensitivity to AT-02 or any of its excipients.
19. Brain MRI performed within 6 months of Screening, or during the Screening period, that shows evidence of any of the following:

    1. Acute or sub-acute hemorrhage.
    2. Prior macrohemorrhage (defined as >1 cm in diameter on T2* sequence or susceptibility-weighted imaging (SWI)) or prior subarachnoid hemorrhage unless it can be documented that the finding is not due to an underlying structural or vascular abnormality (i.e., finding does not suggest participant is at risk of recurrent hemorrhage).
    3. Greater than 4 microhemorrhages (defined as <1 cm in diameter on T2* sequence or SWI).
    4. Cortical infarct (defined as >1.5 cm in diameter; irrespective of anatomic location).
    5. >1 lacunar infarct (defined as <1.5 cm in diameter).
    6. Superficial siderosis.
    7. Any finding that, in the opinion of the Investigator, might pose a risk to the participant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence, frequency, and severity of Treatment-emergent adverse events (TEAEs) as assessed National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) | Up to 112 weeks
To assess the safety and tolerability of AT-02 through change from baseline in clinical laboratory results | Up to 112 weeks

SECONDARY OUTCOMES:
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: maximum observed concentration of AT-02 (Cmax)
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: time to maximum observed AT-02 concentration (Tmax)
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: AUClast
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: AUCinf
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: volume of distribution at steady state (Vss)
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: total body clearance (CL) of AT-02
To assess PK of AT-02 during long-term administration | Up to 112 weeks
  Parameter: AT-02 half-life (t½)
Incidence of treatment-emergent Anti-drug antibodies (ADAs) | Up to 112 weeks
  The number and percentage of subjects who develop detectable ADA will be summarized by dose cohort.
To evaluate the clinical efficacy of AT-02 during long-term administration through change from baseline in biomarkers | Up to 112 weeks
  Biomarkers include serum N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
To evaluate the clinical efficacy of AT-02 during long-term administration through change from baseline in biomarkers | Up to 112 weeks
  Biomarkers include serum High-sensitivity cardiac troponin T (hsTnT)
To evaluate the clinical efficacy of AT-02 during long-term administration through change from baseline in biomarkers | Up to 112 weeks
  Biomarkers include serum Urine albumin creatinine ratio (UACR)
Serial cardiac magnetic resonance assessments of systemic amyloidosis | Up to 112 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kansas City, Kansas City, Kansas
  - Cleveland Clinic, Cleveland, Ohio
  - OHSU (Oregon Health & Science University), Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania